CLINICAL TRIAL: NCT06153446
Title: Comparing Diagnostic Accuracy of Synovasure Comprehensive Synovial Fluid Testing to Clinical Guidelines for the Diagnosis of Periprosthetic Joint Infection
Brief Title: Infection Consortium Study#1
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: DTU2023-02DI
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: PJI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- CDL PJI Database: Patients tested for PJI through the PJI Panel at CD Laboratories (CDL)
  Interventions: Diagnostic Test: Synovasure® Comprehensive Infection Panel

INTERVENTIONS:
Diagnostic Test: Synovasure® Comprehensive Infection Panel — The Synovasure Comprehensive PJI Test Panel (PJI Panel) is a laboratory-developed test (LDT) panel (CD Laboratories, CLIA Registration No.: 21D0216863) intended to aid the diagnosis of PJI.

SUMMARY:
In this study, the Sponsor wants to evaluate the performance and accuracy of the PJI Panel compared to the currently used multiple-criterion scoring systems for the diagnosis of PJI.

DETAILED DESCRIPTION:
This study aims to evaluate the performance and accuracy of the PJI Panel compared to the currently used multiple-criterion scoring systems for the diagnosis of PJI and will be executed as a retrospective review of existing data.

The Synovasure R&D database consists of PJI Panel test results digitally transferred from the instruments to a laboratory information system (LIS), (CGM LabDAQ, CompuGroup Medical, Phoenix, AZ), which has high data-integrity architecture built on an industry standard ACID (atomicity, consistency, isolation, durability) compliant relational database management system (RDBMS), Microsoft SQL Server. These PJI Panel data come from SF samples submitted to CDL from various clinics and hospitals for clinical diagnostic testing between 2013 and 2022 (CD Laboratories, Towson, MD). The data are deidentified in accordance with an existing IRB approval (WCG-IRB #20150222). The deidentified data includes the institution, ordering physician information, anatomical location of the aspiration, number of days from aspiration to receipt of the sample at the lab, age, gender, and results of comprehensive infection testing including: specimen integrity (red blood cells (RBC) and absorbance at 280 nm (A280)), AD, HNE, CRP, WBC, %PMN, MID Panel, and SF-Cx.

The Synovasure R&D database will be submitted to an exclusion/inclusion screening process to target samples for inclusion in this research activity. Subsequently, samples collected between 2017 and 2022 will be randomly selected for inclusion in this study. Classification of positive and negative samples will be according to the criteria for diagnosis of PJI using Synovasure Comprehensive PJI Synovial Fluid Panel as defined in Table 1. Only samples classified as Infected (positive) and Not Infected (negative) will be qualified for further enrichment.

Case report forms will be completed with data obtained through in-person or remote review of hospital and/or physician office records to enrich the PJI Panel database with the elements included in the 2011 MSIS, 2013 ICM, 2018 New Definition of PJI, 2018 ICM, and 2021 EBJIS definitions of PJI.

ELIGIBILITY:
Inclusion Criteria:

* Samples included in the Synovasure R&D database from patients tested for PJI through the PJI Panel at CDL.

Exclusion Criteria:

* From Synovasure Database

  * Samples not submitted to CDL for PJI testing
  * Samples submitted to CDL from Institutions not participating in this study
  * Samples designated as being from anatomical locations other than "left hip", "left knee", "right hip", "right knee
  * Samples without SF-Cx results
  * Samples without SF-CRP results
  * Samples without AD results
  * Samples without WBC results
  * Samples without %PMN results
  * Samples with RBCs ≥ 1 million
  * Samples not meeting A280 specification for integrity: Remove A280 < 0.342 and A280 > 1.19
  * Samples received more than four (4) days after aspiration
  * Patient age < 18 From Institutional Medical Record
  * Patient who did not undergo surgical interventions after PJI Panel Testing
  * Synovasure testing performed less than 6 weeks after index surgery
  * Evidence of sinus tract communicating with the joint
  * Samples aspirated from patients using a spacer at the time of aspiration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient tested for PJI through the PJI Panel at CD Laboratories (CDL).
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2023-12-10 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Positive/Negative Percent Agreement between PJI RISC Panel and Clinical Guidelines | 1 year
  The primary endpoint of this study is the rate of agreement (positive and negative) for the diagnosis of PJI between the PJI Panel and the previous and current clinical guidelines.

SECONDARY OUTCOMES:
Positive/Negative Predictive Value of PJI RISC Panel | 1 year
  The secondary endpoint is defined by the estimate of positive predictive value (PPV) and negative predictive value (NPV) of the PJI Panel compared to the previous and current clinical guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Yale Fillingham, M.D., Principal Investigator — Rothman Institute; Paul Edwards, M.D., Principal Investigator — Bowen Hefley Orthopedics
Locations (1):
- Rothman Orthopedic Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided